CLINICAL TRIAL: NCT02244749
Title: Role of Metabolic Enzymes in Non-Melanoma Skin Cancer: Potential for Informative Biomarkers and Therapeutic Targets
Brief Title: Role of Metabolic Enzymes in Non-Melanoma Skin Cancer
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Chao Family Comprehensive Cancer Center (Other); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kirsten Kelly, M.D., Professor of Dermatology and Surgery, University of California, Irvine
Other Study IDs: 20107851; SEED Grant 405181-66496 (Other: NCI)
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- skin specimen: skin specimen
  Interventions: Other: skin specimen

INTERVENTIONS:
Other: skin specimen — skin specimen

SUMMARY:
The researcher can proved that certain compounds play an important role in the prevention of skin cancer. Researcher can use specific compounds, which classified as metabolic enzymes, and lower concentrations and complete absent in skin cancer cells. Researcher can biopsies of normal skin and precancerous or cancerous lesions, and can compare the concentrations of these compounds to determine the difference between the two areas. The result can lead to further understanding of skin cancers and pre-cancers. Because skin cancers and pre-cancers are so common, any knowledge would be very useful for many people in the future and may be used for development of future treatments or prevention strategies.

DETAILED DESCRIPTION:
Biopsy procedure will be done at the Beckman Laser Institute or at the Dermatology Clinic Gottschalk Medical Plaza, of University of California, Irvine. Standard procedure of punch biopsy will be done in the areas determined by the physician researchers. The normal skin biopsy will be obtained from an area of skin without any suspicious lesions located on an area of the body. Biopsy specimens will be stored frozen at Beckman Laser Institute chemistry-lab for research and will be assigned with subject ID number, there will be no personnel health information attach to the skin specimens. There will be no cost to the subject or their insurer for participation in this study, except in the specific scenario of a suspected skin cancer that would undergo biopsy regardless of participation in this study. The time commitment for each subject is approximately 1 hour for each set of biopsies.

Researchers can test the hypothesis that expression of key metabolic enzymes is reduced and/or lost during skin cancer progression. Total ribonucleic acid, a single-stranded biologic molecule involved in gene transcription, regulation, and translation, can be isolated from biopsied skin specimens. Quantitative Real-Time can be performed to determine the expression levels of several key metabolic enzymes.

Metabolic enzymes regulate several vital signaling pathways in the human body. Some examples include hormone and bioactive lipid regulation. Aberrant regulation of these signaling pathways can lead to human diseases including cancer.

Recent evidence has shown that metabolic enzyme call UGT in the genes call UDP-glucuronosyltransferases were shown to have significantly reduced expression in breast tumors compared with normal breast tissue from the same patients This observed loss of expression is hypothesized to be causal as these two enzymes are responsible for estrogen metabolism.

However, relatively little is known about metabolic enzymes and skin cancer. We have preliminary data that UGT enzyme expression is lost during melanoma progression which allows deregulated lipoxygenase signaling.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female are age18 years and older
* Have normal skin and a skin lesion of interest
* Willing to have skin biopsies on those areas

Exclusion Criteria:

* Male or Female are under 18 years of age
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine Medical Cencal
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
expression levels of metabolic enzymes in normal skin versus precancerous lesions or skin cancer | 1 month
  Overall, compare normal skin versus precancerous lesions or skin cancer from the same individual. Paired tests of samples are selected from the same subjects.
  * 10 actinic keratosis samples,
  * 10 basal cell carcinoma samples
  * 20 squamous cell carcinoma samples
  * Normal skin control biopsy from the same subject will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute, UCI
Locations (2):
- United States (2):
  - Beckman Laser Institute, Irvine, California
  - Gottschalk Medical Plaza, 1 Medical Plaza Drive, Irvine, California